CLINICAL TRIAL: NCT05836610
Title: Hydrocortisone Therapy Optimization During Hypothermia Treatment in Asphyxiated Neonates - a Pharmacokinetic Study
Brief Title: Hydrocortisone Therapy Optimization During Hypothermia Treatment in Asphyxiated Neonates
Acronym: UniCort
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Kata Kovacs, Assistant lecturer, Semmelweis University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SU-Ped-AsphCort 002
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Hypoxic-Ischemic Encephalopathy; Asphyxia; Hypotension; Circulatory Failure Neonatal
Keywords: Hypothermia treatment; Relative adrenal insufficiency; Hydrocortisone supplementation; Hydrocortisone pharmacokinetics; Hypoxic-Ischemic Encephalopathy; Asphyxia
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Asphyxia; Hypotension | interventions — Hydrocortisone; hydrocortisone hemisuccinate

STUDY DESIGN:
Intervention Model Description: Pharmacokinetic analysis of the standard dose hydrocortisone therapy (0.5 mg/kg/6 hours) during hypothermia treatment, then compare the effects of the modified dose hydrocortisone therapy which will be determined based on the pharmacokinetic results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard dose hydrocortisone (Active Comparator): The standard dose of hydrocortisone therapy in neonates for hypotension is 0.5 mg/kg every 6 hours.
  Interventions: Drug: Hydrocortisone
- Modified dose hydrocortisone (Active Comparator): The modified dose of hydrocortisone therapy will be determined based on the pharmacokinetic results.
  Interventions: Drug: Hydrocortisone

INTERVENTIONS:
Drug: Hydrocortisone — intravenous bolus hydrocortisone therapy during hypothermia treatment
  Other Names: Solu-Cortef

SUMMARY:
This is a prospective, single center, pharmacokinetic study of intravenous hydrocortisone therapy for systemic low blood pressure during hypothermia treatment in asphyxiated newborns. Patients will be allocated to hydrocortisone supplementation while receiving conventional inotropic therapy as needed.

The hypothesis is that a detailed study of hydrocortisone pharmacokinetics during therapeutic hypothermia would help to personalize steroid supplementation in asphyxiated neonates. As the overall metabolic rate decreases with lower body temperature, drug metabolism is likely to be reduced as well, and lower doses, or less frequent dosing will be sufficient to achieve the targeted steroid range and biological effects in asphyxiated neonates with relative adrenal insufficiency. Thus, the investigators are planning to measure initial, baseline serum cortisol levels and serial serum cortisol levels after hydrocortisone supplementation in cooled asphyxiated neonates.

DETAILED DESCRIPTION:
The ultimate goal of the present study, is to describe a new approach of more personalized and safe care to infants with birth asphyxia and hemodynamic instability.

Asphyxiated infants often present with multiorgan failure and low blood pressure. Therapeutic hypothermia, the standard of care, could worsen hemodynamic instability; therefore, treatment of cardiovascular impairment represents a major challenge in this clinical setting. An association was previously described between hypotension and low serum cortisol values in this patient population, and it was suggested that relative adrenal insufficiency (RAI) is an important factor in the circulatory compromise of these patients. In the "CORTISoL" clinical trial, it was also demonstrated that low-dose hydrocortisone therapy was effective in the treatment of cardiovascular impairment in asphyxiated neonates; however, some gaps remain in the knowledge on optimal dosing. Importantly, steroid therapy should be administered at the lowest effective dose and for the shortest possible duration in this vulnerable population.

In the current pharmacokinetic study, the investigators propose a stepwise approach to more detailed understanding of RAI and hydrocortisone pharmacokinetics in asphyxiated neonates. The findings would certainly aid clinical decision-making and allow for more personalized therapeutic interventions for the treatment of hemodynamic instability.

ELIGIBILITY:
Inclusion Criteria:

* gestational age ≥ 36 weeks
* provision of whole-body hypothermia treatment (as described by Azzopardi et al.)
* presence of systemic hypotension (defined as a mean arterial pressure less than the gestational age in weeks)
* indication for hydrocortisone treatment during hypothermia by the attending physician
* indwelling arterial catheter to take blood samples without additional painful punctures: umbilical arterial catheter or peripheral arterial catheter
* written informed parental consent

Exclusion Criteria:

* infants who are expected to be > 6 hours of age (not suitable for cooling)
* critical congenital abnormalities
* genetic disease
* signed informed consent is unavailable

Max Age: 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2021-09-21 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Mean blood pressure increase | 2 hours
  5 mmHg increase in mean arterial blood pressure after drug administration

SECONDARY OUTCOMES:
Cardiovascular management | 72 hours
  Length, cumulative and peak dose of inotrope treatment
Presence of relative adrenal insufficiency at baseline | Before hydrocortisone administration within max. 72 hours
  Low serum cortisol level at baseline
MRI outcome | 4-10 days
  Brain injury on MRI examinations
Long term neurodevelopmental outcome | 18-42 month
  Performance on motor and mental scales of Bayley III scales of infant development

OTHER OUTCOMES:
Multiorgan failure | 72 hours
  Presence of multiorgan failure during hypothermia

CONTACTS AND LOCATIONS:
Overall Officials: Kata Kovacs, MD, PhD, Principal Investigator — Semmelweis University; Miklós Szabó, MD, PhD, Study Director — Semmelweis University
Locations (1):
- Semmelweis University Department of Pediatrics (Bókay street Unit), Budapest, Pest County, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Azzopardi DV, Strohm B, Edwards AD, Dyet L, Halliday HL, Juszczak E, Kapellou O, Levene M, Marlow N, Porter E, Thoresen M, Whitelaw A, Brocklehurst P; TOBY Study Group. Moderate hypothermia to treat perinatal asphyxial encephalopathy. N Engl J Med. 2009 Oct 1;361(14):1349-58. doi: 10.1056/NEJMoa0900854. PMID 19797281
- [Background] Kovacs K, Szakmar E, Meder U, Szakacs L, Cseko A, Vatai B, Szabo AJ, McNamara PJ, Szabo M, Jermendy A. A Randomized Controlled Study of Low-Dose Hydrocortisone Versus Placebo in Dopamine-Treated Hypotensive Neonates Undergoing Hypothermia Treatment for Hypoxic-Ischemic Encephalopathy. J Pediatr. 2019 Aug;211:13-19.e3. doi: 10.1016/j.jpeds.2019.04.008. Epub 2019 May 30. PMID 31155392
- [Background] Kovacs K, Szakmar E, Meder U, Cseko A, Szabo AJ, Szabo M, Jermendy A. Serum cortisol levels in asphyxiated infants with hypotension. Early Hum Dev. 2018 May;120:40-45. doi: 10.1016/j.earlhumdev.2018.03.003. Epub 2018 Apr 4. No abstract available. PMID 29626704
- [Background] Watterberg KL. Hydrocortisone Dosing for Hypotension in Newborn Infants: Less Is More. J Pediatr. 2016 Jul;174:23-26.e1. doi: 10.1016/j.jpeds.2016.04.005. Epub 2016 May 4. No abstract available. PMID 27156187
- [Background] Concepcion KR, Zhang L. Corticosteroids and perinatal hypoxic-ischemic brain injury. Drug Discov Today. 2018 Oct;23(10):1718-1732. doi: 10.1016/j.drudis.2018.05.019. Epub 2018 May 17. PMID 29778695
- [Background] Sarkar S, Barks JD. Systemic complications and hypothermia. Semin Fetal Neonatal Med. 2010 Oct;15(5):270-5. doi: 10.1016/j.siny.2010.02.001. Epub 2010 Mar 12. PMID 20227357